CLINICAL TRIAL: NCT01932515
Title: Diagnostic Instruments for Autism in Deaf Children Study
Acronym: DIADS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Leeds and York Partnership NHS Foundation Trust (Other Government)
Collaborators: University of Manchester (Other); Newcastle University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BH120870
Record Dates: First submitted 2013-08-27; First posted 2013-08-30 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Hearing Loss; ASD
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Screening (No Intervention)
  Interventions: Behavioral: A revised screening instrument for use in Deaf children

INTERVENTIONS:
Behavioral: A revised screening instrument for use in Deaf children

SUMMARY:
The trial is in three stages and will translate and validate screening and assessment instruments for use with deaf children.

The first stage is modifying the screening and assessment instruments (ADI-R and ADOS-2) for use with deaf children. This will involve choosing the most promising screening instrument (SRS-2) based on the systematic review and the expertise of a review panel, which contains experts and public and patient involvement (PPI). This phase of the study seeks a wide range of user (parents/ carers and young people) views and experiences about the symptomatology and presentation of deaf children with autism, comparing this to hearing children with autism, and deaf children without autism.

The second stage is to ensure that the newly modified instruments are accessible to deaf children and deaf parents by making any necessary translations from English into British Sign Language. This involves a strict translation and back translation methodology with reiterations until successful translation is achieved.

For stage three in order to ensure that the new questionnaires are successfully identifying children and young people with Autism Spectrum Disorder, the modified instrument will be validated using a 'gold standard'. The current 'gold standard' for the mental health screening of Deaf children is a clinical interview administered by experienced senior multidisciplinary deaf child mental health clinicians.

ELIGIBILITY:
Inclusion Criteria:

For the purposes of this study, children and young people will be recruited if they have a chronological age of ≥18 months old, up to 18 years.

Deaf children will have a hearing loss of at least 40dB

Exclusion Criteria:

This is a pragmatic trial which recognises the frequency and complexity of co-morbidities in children with Autistic Spectrum Disorders (ASD) and deafness. We will therefore not exclude on the basis of co-morbidity in the groups where a diagnosis of ASD already exists, since these tools would be used with this population if adopted more widely in the NHS.

We will not exclude children or young people with language delay as children with ASD may have severe language delay. Families where the parents do not have either a signed language being studied here, or a language in which the ADI-R is available, will not be included.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 325 (Estimated)
Dates: Start 2013-11; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
A validated Autism Spectrum Disorder screening instrument to identify those in need of further assessment from deaf children suspected of ASD, with both English and BSL versions (for deaf parents). | 42 months

SECONDARY OUTCOMES:
A modified version of the Autism Diagnostic Interview Revised (ADIR) validated for use in the assessment of deaf young people; accessible in English and BSL (for hearing and deaf parents to fully participate in assessment). | 42 months

OTHER OUTCOMES:
A modified version of the Autism Diagnostic Observation Schedule (ADOS 2) validated for use with deaf young people in both BSL or English. | 42 months

CONTACTS AND LOCATIONS:
Overall Officials: Barry Wright, Principal Investigator — Leeds and York Partnership NHS Foundation Trust
Locations (1):
- Leeds and York Partnership NHS Foundation Trust, York, North Yorkshire, United Kingdom